CLINICAL TRIAL: NCT04612777
Title: A Trial of "Opening Doors to Recovery" for Persons With Serious Mental Illnesses
Acronym: ODR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Michael Compton, Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7419
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Mental Disorders, Severe; Schizophrenia and Related Disorders; Bipolar Disorder; Depressive Disorder
Keywords: serious mental illness; community navigation
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder | interventions — Case Management

STUDY DESIGN:
Intervention Model Description: Participants will be randomized either to the intervention ("Opening Doors to Recovery") or standard treatment (Intensive Case Management or Case Management)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opening Doors to Recovery (Experimental): Participants will receive services from the team of three ODR navigators: one professional social worker, one navigator who is a family member of someone with SMI, and one peer navigator with lived experience.
  Interventions: Behavioral: Opening Doors to Recovery
- Intensive Case Management or Case Management (Active Comparator): Participants randomized to the control group will either receive standard services of Intensive Case Management or Case Management, depending on the services that are available in their county.
  Interventions: Behavioral: Case Management; Behavioral: Intensive Case Management

INTERVENTIONS:
Behavioral: Opening Doors to Recovery — Opening Doors to Recovery (ODR) was created by a large, collaborative group in southeast Georgia as a recovery-oriented approach that navigates clients into services that may in some cases be fragmented and seemingly inaccessible. The team of three Community Navigation Specialists (CNSs) strives to help clients reduce institutional (e.g., hospital, jail) recidivism and embrace recovery. Their process of community navigation is a broader function than traditional case management as it includes mapping out and connecting clients to all available local resources, which requires being embedded in the community. The work of the CNSs benefits from commitments of diverse collaborative ODR partners, including local treatment providers, law enforcement, employers, and housing programs. Each CNS was expected to meet with the client at home or in community settings at least monthly, with the client having contact with at least one CNS weekly.
  Arms: Opening Doors to Recovery
Behavioral: Case Management — Case Management (CM) services, as defined by the State mental health agency, consist of providing essential environmental support and care coordination to assist the individual with improving his/her functioning, gaining access to necessary services, and creating an environment that promotes recovery as identified in his/her Individual Recovery Plan (IRP). The focus of interventions include assisting the individual with: (1) developing natural supports to promote community integration, (2) identifying service needs, (3) referring and linking to services and resources identified through the service planning process, (4) coordinating services identified on the IRP to maximize service integration and minimize service gaps, and (5) ensuring continued adequacy of the IRP to meet his/her ongoing and changing needs. Contact must be made with the individual ≥2 times per month, at least one of which must be in-person, in a non-clinic setting.
  Arms: Intensive Case Management or Case Management
Behavioral: Intensive Case Management — Intensive Case Management (ICM) is very similar to CM, but four in-person visits are required monthly. Additional contacts may be either face-to-face or via telephone, depending on the individual's needs. At least 60% of total contacts must be face-to-face with the individual, and at least 50% must be delivered in non-clinic/community-based settings. An ICM team includes nine professionals: a licensed clinician, four masters-level clinicians, two bachelors-level clinicians, and two paraprofessionals. The team's maximum case load is 200 in rural settings and 300 in urban settings (22-33 per team member).
  Arms: Intensive Case Management or Case Management

SUMMARY:
Insufficient community-based support after inpatient discharge for persons with serious mental illnesses (SMI) may lead to re-hospitalization, excessive criminal justice involvement, homelessness, and an inability to embrace recovery. In fact, many of these especially vulnerable persons find themselves in a cycle of repeated hospital stays, arrests, and even homelessness, with little support for real recovery. Public mental health systems are struggling to address these problems. Evidence-based, comparatively inexpensive, time-limited community support models are needed to reduce institutional recidivism and facilitate recovery. The Georgia chapter of the National Alliance on Mental Illness (NAMI-GA) developed Opening Doors to Recovery (ODR), and we have collected extensive preliminary data on it. ODR is now being tested in a randomized controlled trial (RCT) taking place in southeast Georgia where ODR was first developed. The primary goals of ODR are to prevent institutional recidivism (i.e., going back into the hospital) and to promote recovery among persons with SMI like schizophrenia and bipolar disorder. The ODR intervention is comprised of several components that work together to address barriers to successful integration into the community among individuals with SMI and repeated inpatient hospitalizations. A team of 3 specially trained "Community Navigation Specialists" (CNSs, also called Navigators) provides intensive, mobile, community support to persons with SMI with a defined history of inpatient recidivism (i.e., repeated hospital stays).

We are carrying out a fully powered trial of ODR in a 7-county catchment area in southeast Georgia, which is an ideal real-world location to carry out the study. During the 5-year study period, we will randomize 240 persons with SMI and a history of ≥2 inpatient stays in the past 12 months to ODR (n=120, followed for 12 months, with a maximum CNS caseload of 40) versus community care in traditional intensive case management or case management (ICM/CM, n=120). Assessments are conducted at baseline (just before hospital discharge), and at 4, 8, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak/read English
* Clinical diagnosis of one of the following: psychotic disorder, bipolar disorder, or major depressive disorder
* Capacity to give informed consent
* Being discharged to one of seven counties served by Gateway Behavioral Health Services
* Being hospitalized on an adult, non-forensics unit at Georgia Regional Hospital at Savannah, the Gateway-Brunswick CSU, or the Savannah CSU (located at Coastal Harbor) for ≥2 nights
* At least one additional prior hospitalization or CSU stay of ≥2 nights within the past 12 months (our definition of "institutional recidivism")
* Inability to complete activities of daily living in at least two of the following areas despite support from caregiver or behavioral health staff (this is a criterion previously established for receiving ICM services):

  1. navigate and self-manage necessary services,
  2. maintain personal hygiene, meet nutritional needs,
  3. care for personal business affairs, obtain or maintain medical, legal, and housing services,
  4. recognize and avoid common dangers or hazards to self and possessions,
  5. perform daily living tasks,
  6. obtain or maintain employment at a self-sustaining level or consistently perform homemaker roles (meal preparation, washing clothes, budgeting, or childcare tasks and responsibilities),
  7. maintain safe living situation (evicted from housing/recent loss of housing/imminent risk of loss of housing)
* Requires assistance with one or more of the following as an indicator of demonstrated ownership and engagement with his/her own illness self-management (this also is a criterion previously established for receiving ICM services): a. Taking prescribed medications b. Following a crisis plan c. Maintaining community integration d. Keeping appointments with needed services which have resulted in the exhibition of specific behaviors that have led to two or more of the following within the past 18 months (hospitalization, incarcerations, homelessness, or use of other crisis services)

Exclusion Criteria:

* Known or suspected intellectual disability, mental retardation, or dementia
* Known or suspected autism-spectrum disorder, organic mental disorder, and/or traumatic brain injury
* Significant medical condition compromising ability to participate (e.g., short of breath, in pain)
* Having taken part in the initial ODR study or being enrolled in any other study.
* Being referred to ACT
* Not having the ability to provide informed consent for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-06-15 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-05-31 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Compton MT, Kelley ME, Anderson S, Ellis S, Graves J, Broussard B, Pauselli L, Zern A, Pope LG, Johnson M, Haynes NL. Opening Doors to Recovery: A Randomized Controlled Trial of a Recovery-Oriented Community Navigation Service for Individuals With Serious Mental Illnesses and Repeated Hospitalizations. J Clin Psychiatry. 2023 Jan 16;84(2):22m14498. doi: 10.4088/JCP.22m14498. PMID 36652687

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Case Management or Case Management: Participants randomized to the control group will either receive standard services of Intensive Case Management or Case Management, depending on the services that are available in their county.
  Case Management (CM) services consist of providing essential environmental support and care coordination to assist the individual with improving his/her functioning, gaining access to necessary services, and creating an environment that promotes recovery as identified in his/her Individual Recovery Plan (IRP). The focus of interventions includes assisting the individual with: (1) developing natural supports to promote community integration, (2) identifying service needs, (3) connecting them to services and resources, (4) coordinating services identified on the IRP to maximize service integration and minimize service gaps, and (5) ensuring continued adequacy of the IRP to meet his/her ongoing and changing needs. Contact must be made with the individual ≥2 times per month, at least one of which must be in-person, in a non-clinic setting.
  Intensive Case Management (ICM) is very similar to CM, but 4 in-person visits are required monthly. At least 60% of contacts must be face-to-face, and at least 50% must be delivered in non-clinic settings. ICM teams include 9 professionals: a licensed clinician, 4 masters-level clinicians, 2 bachelors-level clinicians, and 2 paraprofessionals. The team's maximum caseload is 200 in rural settings and 300 in urban settings (22-33 per team member).
Period: Overall Study
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Started | 117 | 123
4 Months | 109 | 109
8 Months | 106 | 106
Completed | 100 | 100
Not Completed | 17 | 23

BASELINE CHARACTERISTICS:
Groups:
- Intensive Case Management or Case Management: Participants randomized to the control group will either receive standard services of Intensive Case Management or Case Management, depending on the services that are available in their county.
  Case Management (CM) services consist of providing essential environmental support and care coordination to assist the individual with improving his/her functioning, gaining access to necessary services, and creating an environment that promotes recovery as identified in his/her Individual Recovery Plan (IRP). These interventions include assisting the individual with: (1) developing natural supports to promote community integration, (2) identifying service needs, (3) connecting them to services and resources, (4) coordinating services identified on the IRP, and (5) ensuring continued adequacy of the IRP to meet their ongoing and changing needs. Contact must be made with the individual ≥2 times per month, and at least once in-person, in a non-clinic setting.
  Intensive Case Management (ICM) is similar to CM, but 4 in-person visits are required monthly. Additional contacts may be in-person or telephonic. At least 60% of total contacts must be in-person with the individual, and at least 50% must be delivered in non-clinic settings. An ICM team includes 9 professionals: a licensed clinician, 4 masters-level clinicians, 2 bachelors-level clinicians, and 2 paraprofessionals. The team's maximum caseload is 200 in rural settings and 300 in urban settings (22-33 per team member).
- Total: Total of all reporting groups
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management | Total
Number analyzed (Participants) | 117 | 123 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 123 | 240
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.8 (11.8) | 36.0 (11.4) | 35.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 49 | 85
  Male | 81 | 74 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 106 | 112 | 218
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 58 | 114
  White | 55 | 61 | 116
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117 | 123 | 240

OUTCOME MEASURES:

1. Primary Outcome: Number of Inpatient Psychiatric Stays for Intervention and Control Participants
Description: Data on inpatient psychiatric stays will be collected from the Georgia Department of Behavioral Health and Developmental Disabilities, Gateway Behavioral Health Services Crisis Stabilization Unit in Brunswick, Georgia, and Coastal Harbor Crisis Stabilization Unit in Savannah, Georgia.
  Hypothesis A1: ODR participants will have fewer inpatient psychiatric stays during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
Hospitalizations | 1.9 (1.5) | 2.3 (1.8)

2. Primary Outcome: Number of Arrests for Intervention and Control Participants
Description: Participants' Record of Arrest and Prosecution (RAP) sheets will be collected from the Georgia Bureau of Investigation, and data on each participant's arrests during the study period will be extracted.
  Hypothesis B1: ODR participants will have fewer arrests during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Deviation); unit: number of arrests
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
number of arrests | 1.7 (1.1) | 2.0 (1.3)

3. Primary Outcome: Number of Days Hospitalized for Intervention and Control Participants
Description: Data on inpatient psychiatric days will be collected from the Georgia Department of Behavioral Health and Developmental Disabilities, Gateway Behavioral Health Services Crisis Stabilization Unit in Brunswick, Georgia, and Coastal Harbor Crisis Stabilization Unit in Savannah, Georgia.
  Hypothesis A2: ODR participants will have fewer inpatient psychiatric hospital days during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Deviation); unit: days hospitalized
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
days hospitalized | 18.0 (15.1) | 20.7 (27.0)

4. Secondary Outcome: Scores on the Housing Instability Index (HII)
Description: The Housing Instability Index will be administered orally to all study participants during the routine follow-up assessments at 4-months, 8-months, and 12-months. It contains 10 items. The measure was scaled on a scale of 0 to 10 with higher scores indicating greater housing instability. We computed a "change score" representing the participant's change in scores from baseline to 12-months. Group effects are shown as the mean difference (Δ) from baseline to 12 months per group, but estimates are derived from fitted linear slope of change over all data (baseline, 4 months, 8 months, and 12 months).
  Hypothesis C1a: ODR participants will have lesser housing instability during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
units on a scale | -2.97 (0.27) | -2.48 (0.30)

5. Secondary Outcome: Scores on the Housing Satisfaction Scale (HSS)
Description: The Housing Satisfaction Scale (HSS) will be administered orally to all study participants during the routine follow-up assessments at 4-months, 8-months, and 12-months. It contains 19 items covering choice, safety, privacy, and proximity. The measure was scaled on a scale of 1 to 5, with higher scores indicate lesser housing satisfaction. We computed a "change score" representing the participant's change in scores from baseline to 12-months. Group effects are shown as the mean difference (Δ) from baseline to 12 months per group, but estimates are derived from fitted linear slope of change over all data (baseline, 4 months, 8 months, and 12 months).
  Hypothesis C1b: ODR participants will have greater housing satisfaction during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
units on a scale | -0.88 (0.09) | -0.52 (0.10)

6. Secondary Outcome: Scores on the Multnomah Community Ability Scale (MCAS)
Description: At each routine follow-up assessments at 4-months, 8-months, and 12-months, participants will respond to the Multnomah Community Adjustment Scale .It contains 17 items that measure social and community functioning; 5 other items were added. The measure was scaled on a scale of 1 to 5, with higher scores indicate greater community abilities. We computed a "change score" representing the participant's change in scores from baseline to 12-months. Group effects are shown as the mean difference (Δ) from baseline to 12 months per group, but estimates are derived from fitted linear slope of change over all data (baseline, 4 months, 8 months, and 12 months).
  Hypothesis D1a: ODR participants will have greater recovery, based on the scale of community adjustment, during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
units on a scale | 0.47 (0.07) | 0.32 (0.08)

7. Secondary Outcome: Scores on the Maryland Assessment of Recovery in People With Serious Mental Illness (MARS)
Description: At each routine follow-up assessments at 4-months, 8-months, and 12-months, participants will respond to the Maryland Assessment of Recovery in People with Serious Mental Illness. It contains 25 items that measure recovery experiences. The measure was scaled on a scale of 1 to 5, with higher scores indicate greater recovery. We computed a "change score" representing the participant's change in scores from baseline to 12-months. Group effects are shown as the mean difference (Δ) from baseline to 12 months per group, but estimates are derived from fitted linear slope of change over all data (baseline, 4 months, 8 months, and 12 months).
  Hypothesis D1b: ODR participants will have greater recovery, based on the MARS scale, during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
units on a scale | 0.22 (0.08) | 0.05 (0.09)

8. Secondary Outcome: Scores on the Herth Hope Scale (HHS)
Description: At each routine follow-up assessments at 4-months, 8-months, and 12-months, participants will respond to the Herth Hope Scale (HHS). It contains 30 items that measure hope. The measure was scaled on a scale of 1 to 5, with higher scores indicate greater hope. We computed a "change score" representing the participant's change in scores from baseline to 12-months. Group effects are shown as the mean difference (Δ) from baseline to 12 months per group, but estimates are derived from fitted linear slope of change over all data (baseline, 4 months, 8 months, and 12 months).
  Hypothesis D1c: ODR participants will have greater recovery, based on the HHS, during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
units on a scale | 0.24 (0.06) | 0.14 (0.06)

9. Secondary Outcome: Scores on the Empowerment Scale
Description: At each routine follow-up assessments at 4-months, 8-months, and 12-months, participants will respond to the Empowerment Scale. It contains 28 items that measure self-esteem, perceived power, optimism/control over the future, and related constructs. The measure was scaled on a scale of 1 to 4, with higher scores indicate greater empowerment. We computed a "change score" representing the participant's change in scores from baseline to 12-months. Group effects are shown as the mean difference (Δ) from baseline to 12 months per group, but estimates are derived from fitted linear slope of change over all data (baseline, 4 months, 8 months, and 12 months).
  Hypothesis D1d: ODR participants will have greater recovery, based on the Empowerment Scale, during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
units on a scale | 0.11 (0.03) | 0.00 (0.03)

10. Secondary Outcome: Scores on the Community Navigation Abilities Scale (CNAS)
Description: At each routine follow-up assessments at 4-months, 8-months, and 12-months, participants will respond to the Community Navigation Abilities Scale (CNAS). It contains 21 items that measure community navigation abilities. The measure was scaled on a scale of 1 to 7, with higher scores indicate greater community navigation abilities. We computed a "change score" representing the participant's change in scores from baseline to 12-months. Group effects are shown as the mean difference (Δ) from baseline to 12 months per group, but estimates are derived from fitted linear slope of change over all data (baseline, 4 months, 8 months, and 12 months).
  Hypothesis D1e: ODR participants will have greater recovery, based on the CNAS, during a 12-month period compared to participants in ICM/CM.
Time Frame: 12 months of study enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
Number analyzed (Participants) | 117 | 123
units on a scale | 1.15 (0.13) | 0.75 (0.14)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Consistent with clinicicaltrials.gov definitions.
Arm/Group | Opening Doors to Recovery | Intensive Case Management or Case Management
All-Cause Mortality (participants affected / at risk) | 0/117 | 3/123
Serious Adverse Events (participants affected / at risk) | 1/117 | 1/123
Other Adverse Events (participants affected / at risk) | 0/117 | 0/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opening Doors to Recovery (N=117) | Intensive Case Management or Case Management (N=123)
Psychiatric symptom exacerbation (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT04612777/Prot_SAP_000.pdf